CLINICAL TRIAL: NCT05653414
Title: Interest of a Short Early Psychological Care in Women With Miscarriage: a Controlled Randomized Study
Brief Title: Interest of a Short Early Psychological Care in Women With Miscarriage
Acronym: MisTher
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022_RIPH_003_MisTher
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2022-12

CONDITIONS: Miscarriage
Keywords: Miscarriage; Psychological care; Anxiety; Depression; Post traumatic stress disorder
MeSH Terms: conditions — Abortion, Spontaneous; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "short early psychological care" group (Experimental): Women with short early psychological care associated with encouragement of early support consultation with generalist practitioner or midwife
  Interventions: Other: short early psychological care associated with encouragement of early support consultation with generalist practitioner or midwife
- "control" group (Active Comparator): Women with encouragement of early support consultation with generalist practitioner or midwife
  Interventions: Other: encouragement of early support consultation with generalist practitioner or midwife

INTERVENTIONS:
Other: short early psychological care associated with encouragement of early support consultation with generalist practitioner or midwife — 4 consultations with a psychologist over 2 months maximum
  Arms: "short early psychological care" group
Other: encouragement of early support consultation with generalist practitioner or midwife — encouragement of early support consultation with generalist practitioner or midwife
  Arms: "control" group

SUMMARY:
Miscarriage is a very common complication of pregnancy, accounting for 15.3% (95% CI 12.5-18.7%) of diagnosed pregnancies. Miscarriage would affect one in ten women during her lifetime. Worldwide, 23 million miscarriages occur annually.

Because of its frequency, miscarriage isoften considered as trivial event by caregivers. Still, miscarriage can be a traumatic event. Literature is consistent on the psychological morbidity associated with miscarriage. Anxiety, depression, post-traumatic stress have been studied in women after miscarriage. Cohort studies and clinical trials suggest that psychological and supportive interventions performed in women after miscarriage may improve women's psychological well-being and reduce miscarriage complications in subsequent pregnancies. However, to date, the literature is considered insufficient on the psychological care of women after a miscarriage.

DETAILED DESCRIPTION:
The aim of the study will be to evaluate the interest of a short early psychological care in women with miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* women with an early miscarriage (defined by a spontaneous termination of pregnancy before the 14th week of amenorrhea)
* women aged more than 18
* women agreeing to participate in the study (signing the informed consent form).

Exclusion Criteria:

* ectopic pregnancy
* molar pregnancy
* women with recurrent miscarriages
* women less than 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 932 (Estimated)
Dates: Start 2023-05-30 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
anxiety | Month 3
  Anxiety will be evaluated using the Scale Trait Anxiety Inventory version Y (STAI-Y-A). The STAI Form Y-A consists of a set of twenty item sonly focus on the psychological and not the somatic aspects of anxiety. The STAI Form Y-A is a self-reported questionnaire. Each item is scored from 1 to 4 and a sum score of all items is computed. Higher score indicates greater anxiety. Presence of anxiety will be defined by a score greater than or equal to 46.

SECONDARY OUTCOMES:
depression | month 3
  depression will be evaluated using Beck Depression Inventory - Second Edition (BDI-II). The BDI-II is a self-reported index of depressive symptoms experienced in the past 2 weeks. The questionnaire includes 21 items of depression symptoms and attitude that the subjects must answer on a 4-point scale from 0 to 3 (0 = not at all bothered; 3 = severely bothered). The minimum score in this questionnaire is 0 and the maximum is 63. Total score indicates that depression is minimal (from 0 to 11 points), mild (from 12 to 19 points), moderate (from 20 to 35 points), or severe (from 36 to 63 points). Presence of depression will be defined by a score greater than or equal to 19.
anxiety | month 6
  Anxiety will be evaluated using the Scale Trait Anxiety Inventory version Y (STAI-Y-A). The STAI Form Y-A consists of a set of twenty item sonly focus on the psychological and not the somatic aspects of anxiety. The STAI Form Y-A is a self-reported questionnaire. Each item is scored from 1 to 4 and a sum score of all items is computed. Higher score indicates greater anxiety. Presence of anxiety will be defined by a score greater than or equal to 46.
depression | month 6
  depression will be evaluated using Beck Depression Inventory - Second Edition (BDI-II). The BDI-II is a self-reported index of depressive symptoms experienced in the past 2 weeks. The questionnaire includes 21 items of depression symptoms and attitude that the subjects must answer on a 4-point scale from 0 to 3 (0 = not at all bothered; 3 = severely bothered). The minimum score in this questionnaire is 0 and the maximum is 63. Total score indicates that depression is minimal (from 0 to 11 points), mild (from 12 to 19 points), moderate (from 20 to 35 points), or severe (from 36 to 63 points). Presence of depression will be defined by a score greater than or equal to 19.

REFERENCES:
- [Derived] Barbe C, Boiteux-Chabrier M, Charillon E, Bouazzi L, Maheas C, Merabet F, Graesslin O, Auer J, Hammami S, Rolland AC, Hurtaud A. Utility of early, short psychological care for women who experience early miscarriage: protocol for the randomized, controlled MisTher trial. BMC Psychol. 2023 Nov 3;11(1):368. doi: 10.1186/s40359-023-01421-x. PMID 37924101